CLINICAL TRIAL: NCT05251870
Title: Tolerogenic Dendritic Cell Therapy for Rheumatoid Arthritis: the TOLERANT Trial
Brief Title: Tolerogenic Dendritic Cell Therapy for Rheumatoid Arthritis
Acronym: TOLERANT
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: UMC Utrecht (Other)
Collaborators: Radboud University Medical Center (Other); Utrecht University (Other); Trajectum Pharma B.V. (Unknown); Dutch Arthritis Association (Industry); ZonMw: The Netherlands Organisation for Health Research and Development (Other); Health Holland (Other)
Responsible Party: Principal Investigator, Jacob M van Laar, Professor of Rheumatology, UMC Utrecht
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NL71296.000.20; 2019-003620-20 (EudraCT Number)
Record Dates: First submitted 2021-12-21; First posted 2022-02-23 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Tolerogenic Dendritic Cells
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intranodal TolDCB29 (low dose) (Experimental): Two administrations of 5 million autologous mature tolerogenic monocyte-derived Dendritic Cells loaded with the B29 peptide of HSP70 (TolDCB29). This cohort will consist of three patients.
  Interventions: Drug: autologous mature tolerogenic monocyte-derived Dendritic Cells loaded with the B29 peptide of HSP70
- Intranodal TolDCB29 (intermediate dose) (Experimental): Two administrations of 10 million autologous mature tolerogenic monocyte-derived Dendritic Cells loaded with the B29 peptide of HSP70 (TolDCB29). This cohort will consist of three patients.
  Interventions: Drug: autologous mature tolerogenic monocyte-derived Dendritic Cells loaded with the B29 peptide of HSP70
- Intranodal TolDCB29 (high dose) (Experimental): Two administrations of 15 million autologous mature tolerogenic monocyte-derived Dendritic Cells loaded with the B29 peptide of HSP70 (TolDCB29). This cohort will consist of three patients.
  Interventions: Drug: autologous mature tolerogenic monocyte-derived Dendritic Cells loaded with the B29 peptide of HSP70
- Intranodal TolDCB29 (recommended dose) (Experimental): Two administrations of the recommended dose of autologous mature tolerogenic monocyte-derived Dendritic Cells loaded with the B29 peptide of HSP70 (TolDCB29). The recommended dose will be advised by the data safety monitoring board after data review of the first three arms. This cohort will consist of nine patients.
  Interventions: Drug: autologous mature tolerogenic monocyte-derived Dendritic Cells loaded with the B29 peptide of HSP70

INTERVENTIONS:
Drug: autologous mature tolerogenic monocyte-derived Dendritic Cells loaded with the B29 peptide of HSP70 — Intranodal administration into an inguinal lymphnode. Two administrations at the same injection site with a four week interval.
  Other Names: TolDCB29

SUMMARY:
Rationale: In rheumatoid arthritis, immune cells cause joint inflammation and destruction in response to autoantigens. Immunosuppressive therapies offer relief but fail to induce tolerance to autoantigens. Injection of antigen-loaded tolerogenic dendritic cells induces immune tolerance and ameliorates disease in arthritis models. The investigators hypothesize that dendritic cell therapy with TolDCB29 is safe and induces immune tolerance in rheumatoid arthritis patients.

Objective: The aim of the study is to demonstrate the safety and feasibility of intranodal TolDCB29 administration. Secondary objectives are the characterization of B29-peptide specific immune reactivity in response to TolDCB29 treatment and the evaluation of the effect of the treatment on disease activity.

Study design: Phase I/II, open-label, dose-escalation clinical trial. Study population: Adult patients (>18 years) with rheumatoid arthritis in remission or low disease activity while on disease modifying anti-rheumatic drugs (DMARD) will be included. Any combination and dose of DMARD is allowed, with exception of Janus kinase inhibitors. Concomitant use of a low dose of prednisone (7.5 mg per day or below) is allowed. Medication should be stable for at least twelve weeks. 18 patients will undergo the experimental treatment.

Intervention: Study participants will receive two intranodal injections with the TolDCB29 product with a four-week interval. During the first phase of the study dose escalation is performed, in which the first group (n=3) receives two "low dose" injections, the second group (n=3) receives two "intermediate dose" injections, and the third group (n=3) receives two "high dose" injections. During the second phase, a fourth group (n=9) will receive the highest dosage without attributable serious adverse events thus far.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of rheumatoid arthritis (RA) according to the criteria which were valid at time of diagnosis (i.e. 1987 Rheumatoid Arthritis Classification or 2010 American College of Rheumatology/EULAR RA Classification Criteria)
* Stable dose, for at least 12 weeks, of any combination of disease-modifying antirheumatic drugs and glucocorticoids (maximum of 7.5 mg per day), with exception of those drugs that are part of the exclusion criteria.
* Disease in remission or in low disease activity for at least 12 weeks (disease activity score of 28 joints < 3.2)
* Able and willing to give informed consent and to comply with the study protocol

Exclusion Criteria:

* Intramuscular or intra-articular glucocorticoid injection during 12 weeks prior to inclusion
* Use of JAK inhibitors
* Active or chronic infection (except fungal nail infection)
* Infection requiring hospitalization or IV antibiotics within 6 weeks of baseline
* Immunization with live vaccine within 6 weeks of baseline
* History of malignancy (except treated basal cell carcinoma of skin)
* Use of other investigational medicinal products within 30 days prior to study entry
* Major surgery within 8 weeks of baseline or planned within 12 weeks from baseline
* Pregnancy, or women planning to become pregnant within the study period, or women who are breast feeding
* Hb<6 mmol/L; neutrophils< 2.00 x10^9/L; platelets <150x10^9/L; alanine aminotransferase or alkaline phosphatase>2x upper limit of normal; renal insufficiency (clearance < 60 ml/min) at screening visit
* Poor venous access or medical condition precluding leukapheresis
* Serious or unstable co-morbidity deemed unsuitable by PI, e.g. chronic obstructive pulmonary disease, cardiac failure
* Individuals of child bearing potential unwilling to use adequate contraception for duration the of study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-08-17 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Safety as assessed by the occurrence and severity of adverse events | 34 weeks
  The occurrence and severity of adverse events will be recorded, including the occurrence of disease flares.
Quantity of good manufacturing practices (GMP)-grade TolDCB29 released according to Quality Control. | 34 weeks
  Number of TolDCB29 cells (millions of cells) per patient that were released according to the quality control standards of the IMPD.
Occurrence of out of specification (OOS) products. | 34 weeks
  Number of occurrences that out of specification TolDCB29 products were generated during manufacturing and/or reconsitution.

SECONDARY OUTCOMES:
Changes in leukocyte numbers | 34 weeks
Changes in CD4+ T lymphocytes subset frequencies | 34 weeks
Lymphocyte proliferation to HSP70/B29 peptide | 34 weeks

OTHER OUTCOMES:
Disease activity of 28 joints (DAS28) | 34 weeks
  Score ranges 0 - 9.4. Higher score means higher disease activity
Quality of life (EQ-5D-5L) | 34 weeks
  Score ranges from less than 0 to 1. In this score, 0 represents a health state equivalent to death and 1 represents full health.
Mean functional ability (HAQ) | 34 weeks
  Score ranges 0 - 3.0 in 0.1 increments. Higher scores indicate worse function and greater disability.
Autoantibody levels | 34 weeks
  Blood autoantibody levels in Units/mL

CONTACTS AND LOCATIONS:
Overall Officials: Jacob M van Laar, MD, PhD, Principal Investigator — UMC Utrecht; Arie J Stoppelenburg, PhD, Study Director — UMC Utrecht
Locations (3):
- Netherlands (3):
  - Radboud University Medical Centre, Nijmegen
  - University Medical Centre Utrecht, Utrecht
  - Utrecht University, Utrecht

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Stoppelenburg AJ, Schreibelt G, Koeneman B, Welsing P, Breman EJ, Lammers L, de Goede A, Duiveman-de Boer T, van Eden W, Leufkens P, de Vries IJM, Broere F, van Laar JM. Design of TOLERANT: phase I/II safety assessment of intranodal administration of HSP70/mB29a self-peptide antigen-loaded autologous tolerogenic dendritic cells in patients with rheumatoid arthritis. BMJ Open. 2024 Sep 12;14(9):e078231. doi: 10.1136/bmjopen-2023-078231. PMID 39266308